CLINICAL TRIAL: NCT06072196
Title: Novel Hormonal Therapies (NHTs) for the Treatment of Metastatic Castration-sensitive Prostate Cancer (mCSPC) in the Medicare Population
Brief Title: A Study to Learn About Novel Hormonal Therapies in People With Metastatic Castration-Sensitive Prostate Cancer (mCSPC)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C3431049; NCT06072196 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms
Keywords: metastatic castration-sensitive prostate cancer; mCSPC; metastatic hormone-sensitive prostate cancer; mHSPC; enzalutamide; abiraterone; treatment duration
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; apalutamide; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novel hormonal therapy cohort: Patients initiating novel hormonal therapy (abiraterone, apalutamide or enzalutamide) for mCSPC
  Interventions: Drug: Novel hormonal therapy

INTERVENTIONS:
Drug: Novel hormonal therapy — As provided in real-world setting
  Other Names: Abiraterone (Yonsa, Zytiga); Apalutamide (Erleada); Enzalutamide (Xtandi)

SUMMARY:
The purpose of this study is to learn about how long novel hormonal therapies are taken by men to treat mCSPC. Novel hormonal therapies in this study include study medicines abiraterone, apalutamide, and enzalutamide.

Prostate cancer is one of the most common cancers in men. The prostate is a gland in the male body that helps make semen. Metastatic cancer is a cancer that has spread to other parts of the body. Castration-sensitive prostate cancer means the cancer is being controlled by keeping the testosterone levels as low as would be expected if the testicles were removed by surgery.

This is a real-world study, not a clinical trial. This means that researchers will look at what happens when men receive the treatments prescribed by their own doctor as part of their usual healthcare treatment. In this study, researchers will use insurance claim information from Medicare claims data.

The study will include patients' information from the database for men who:

* Were identified to have mCSPC.
* Started treatment with novel hormonal therapy (index date) for mCSPC.
* Were 65 years of age or older one year before index date.

Men in this study will be taking novel hormonal therapy for treatment of their mCSPC. We will describe how long men take novel hormonal therapy. This study will use patient information from insurance claims. It will take information one year before start of novel hormonal treatment until the end of insurance period or until information is available.

ELIGIBILITY:
Inclusion Criteria:

* Male with ≥ 1 diagnosis claim for prostate cancer
* Have documented secondary metastasis code on or after the initial prostate cancer diagnosis
* Have initiated novel hormonal therapy (abiraterone, apalutamide, or enzalutamide) within 30 days prior to the metastasis date or on or after the metastasis date. The initiation date of the earliest novel hormonal therapy will be defined as the index date.
* Have a claim for androgen deprivation therapy (ADT) within 90 days prior to or within 30 days after the index date
* ≥65 years old 12 months prior to the index date
* Continuous enrollment in Medicare Parts A, B, and D for ≥12 months prior to the index date and ≥6 months following the index date (unless death)

Exclusion Criteria:

* Claims indicating ≥8 weeks of continuous ADT use between 90 and 365 days prior to the index date, which may indicate castration-resistance
* Received chemotherapy, novel hormonal therapy, radium-223, PARP inhibitor, immunotherapy, or surgical castration prior to the index date
* Had a prior history of other cancers

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men with metastatic castration-sensitive prostate cancer who initiated novel hormonal therapy (abiraterone, apalutamide, or enzalutamide) and met eligibility criteria will be included in the study. Patients will be identified from the 100% Fee-For-Service Medicare claims data.
Sampling Method: Non-Probability Sample
Enrollment: 3017 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3431049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for eligible participants with metastatic castration-sensitive prostate cancer (mCSPC), who initiated a novel hormonal therapy (NHT) [abiraterone or apalutamide or enzalutamide] and had its claim from 01-Jan-2020 to 31-Dec-2021 (index window) were retrieved from existing administrative data from Original Medicare.
Pre-assignment Details: Retrospective data were retrieved and evaluated per objectives of this observational study from 04-Oct-2023 to 18-Dec-2024 (approximately 1.2 years).
Groups:
- Novel Hormonal Therapy: Participants diagnosed with mCSPC and who initiated a NHT (abiraterone, apalutamide or enzalutamide) in real world setting under routine clinical practice were included. Data from these participants were observed retrospectively. No intervention was administered during this study.
Period: Overall Study
Arm/Group | Novel Hormonal Therapy
Started | 3017
Completed | 3017
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants who met inclusion/exclusion criteria, whose data was retrieved and observed in the study.
Arm/Group | Novel Hormonal Therapy
Number analyzed (Participants) | 3017
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.0 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3017
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: Non-Hispanic White | 2,475
  Race/Ethnicity, Customized: Black or African American | 246
  Race/Ethnicity, Customized: Asian/Pacific Islander | 76
  Race/Ethnicity, Customized: Hispanic | 96
  Race/Ethnicity, Customized: Other/Unknown | 124

OUTCOME MEASURES:

1. Primary Outcome: Duration of NHT Treatment
Description: Treatment duration was defined as the time from the initial claim date of NHT (abiraterone, apalutamide, or enzalutamide) until the end of observation for any of the following reasons: (i) end of data availability (December 31, 2022), (ii) participant's date of death, (iii) day before a treatment switch, (iv) day of treatment discontinuation (a 90-day gap in days supply was considered as discontinuation). Retrospective retrieved data collected was evaluated for approximately 1.2 years of this study. Kaplan-Meier method was used for estimation.
Time Frame: 2 years (retrospective data observation duration)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Novel Hormonal Therapy
Number analyzed (Participants) | 3017
Months | 11.9 [11.4 to 12.7]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be evaluated for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not planned to be evaluated (thus at risk appears "0").
Arm/Group | Novel Hormonal Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT06072196/Prot_SAP_000.pdf